CLINICAL TRIAL: NCT06423898
Title: Efficacy and Safety of Ampicillin and Ceftriaxone Continuous Infusion Versus Standard Therapy for the Treatment of Enterococcus Faecalis Infective Endocarditis (DOβLEI Study)
Brief Title: Ampicillin and Ceftriaxone for the Treatment of Enterococcus Faecalis Infective Endocarditis.
Acronym: DOBLEI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOBLEI
Record Dates: First submitted 2024-05-13; First posted 2024-05-21 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Endocarditis, Infective
Keywords: Endocarditis, Infective; Enterococcus faecalis; Antibiotics; Outpatient Infusion Therapies; Outpatient Care
MeSH Terms: conditions — Endocarditis | interventions — Ampicillin; Ceftriaxone

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized 1:1 to experimental group (continuous infusion arm) or control group (intermittent infusion arm)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous intravenous antibiotic infusion (Experimental): Ampicillin 12g/24h plus ceftriaxone 4g/12h continuous infusion. The duration of treatment will be 42 days.
  Interventions: Drug: Ampicillin plus ceftriaxone in continuous infusion
- Standard treatment (Active Comparator): Ampicillin 2g/4h plus ceftriaxone 2g/12h intermittent infusion for a minimum of 14 days. Starting on day 14 of treatment, if the patient is discharged from the hospital, the following treatments will be permitted:
  1. Intravenous treatment in TADE programs according to the following regimens:
     1. Ampicillin 2g/4h plus ceftriaxone 2g/12h as an intermittent infusion
     2. Teicoplanin 10-12mg/kg/24h
     3. Daptomycin 10-12mg/kg/24h
     4. Dalbavancin: Initial dose: 2 doses of 1500mg every 2 weeks. Maintenance dose: 1500mg every 15days.
     5. Linezolid: 600mg/12hours
  2. Oral treatment according to the following regimens:
     1. Amoxicillin 1 g/6h + Moxifloxacin 400mg/24h.
     2. Amoxicillin 1 g/6h + Linezolid 600 mg/12h.
     3. Amoxicillin 1 g/6h + Rifampin 600 mg/12h.
     4. Linezolid 600 mg/12h + Moxifloxacin 400mg/24h.
     5. Linezolid 600 mg/12h + Rifampin 600 mg/12h. The duration of treatment will be 42 days
  Interventions: Drug: Ampicillin plus ceftriaxone in intermittent infusion of 14 days, after which the treatment may be changed

INTERVENTIONS:
Drug: Ampicillin plus ceftriaxone in continuous infusion — Continuous intravenous antibiotic infusion during 42 days for Infective Endocarditis
  Other Names: Experimental regimen
  Arms: Continuous intravenous antibiotic infusion
Drug: Ampicillin plus ceftriaxone in intermittent infusion of 14 days, after which the treatment may be changed — Ampicillin plus ceftriaxone as an intermittent infusion for a minimum of 14 days. After, if the patient is discharged from the hospital, the following treatments, until the 42-day treatment period is completed:
  1. Intravenous treatment according to the following regimens:
     Ampicillin plus ceftriaxone as an intermittent infusion, teicoplanin, daptomycin, dalbavancin or linezolid.
  2. Oral treatment according to the following regimens: amoxicillin plus moxifloxacin, amoxicillin plus linezolid, amoxicillin plus rifampin, linezolid plus moxifloxacin or linezolid plus rifampin.
  Other Names: Control regimen
  Arms: Standard treatment

SUMMARY:
Phase IV, open-label, randomized and multicenter clinical trial to prove that patients with Enterococcus faecalis infective endocarditis treated with an antibiotic treatment as a continuous infusion is non-inferior to the standard treatment, usually administered in hospitalized patients.

DETAILED DESCRIPTION:
The aim of the study is to prove that the continuous infusion of antibiotic treatment for the patients with Enterococcus faecalis infective endocarditis is as effective and safe as the standard treatment. The continuous infusion modality of treatment is expected to provide numerous benefits for individual patients, global health, and for the National Health Care System by reducing to hospital stays from 4-6 weeks to approximately 2-3 weeks and hospital-driven complications.

The mortality, rate of serious adverse events, total number of days of antibiotic treatment and days of hospitalization, among others, are included as secondary objectives.

This is a pragmatic study as the number or visits performed for the study are similar to the normal clinical follow-up for this patients. Final contact and final visit for the study will be performed at 365 days after the 42 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Possible or definitive diagnosis of infective endocarditis due to Enterococcus faecalis
* Signed informed consent of patients

Exclusion Criteria:

* Allergy to penicillins or cephalosporins
* Pregnancy and lactation
* Polymicrobial infection including microorganisms different to E. faecalis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical failure | One year after the end of the treatment
  It is defined as follow:
  i) Confirmed recurrence of E. faecalis infective endocarditis, ii) all-cause mortality. A composite primary endpoint has been chosen to include both a very clinically relevant variable and a hard variable such as survival

SECONDARY OUTCOMES:
Therapeutic failure | Up to 12 months after treatment administration
  Number of deaths
Cardiac surgeries | Up to 12 months after treatment administration
  Number of unplanned cardiac surgeries
Readmissions | Up to 12 months after treatment administration
  Number of unplanned readmissions
Adverse events | From randomisation until 30 days after the last dose administration
  Number of medication-related adverse events
Antibiotic treatment days | Up to 12 months after treatment administration
  Number of antibiotic treatment days
Outpatient Parenteral Antimicrobial Therapy | Up to 12 months after treatment administration
  Number of Outpatient Parenteral Antimicrobial Therapy
Healthcare-associated infections | Up to 12 months after treatment administration
  Number of healthcare-associated infections
Recurrence | Up to 12 months after treatment administration
  Number of recurrence of Enterococcus faecalis infective endocarditis
Minimum free serum concentration | Day 14
  Minimum free serum concentration of antibiotics used
Steady-state plasma concentration | Day 14
  Steady-state plasma concentration of antibiotics used
Pharmacokinetic parameters | Day 14
  Volume of distribution, clearance, elimination constant of antibiotics used
Minimum Inhibitory Concentration | Day 14
  Minimum Inhibitory Concentration of ampicillin induced by ceftriaxone in the strains responsible for recurrences and control strains

CONTACTS AND LOCATIONS:
Overall Officials: HUVR Cesar Arístides de Alarcón González, MD-PhD, Principal Investigator — Fundación para la Gestión de la Investigación en Salud de Sevilla
Locations (18):
- Spain (18):
  - Hospital Universitario de Álava, Alava
  - Hospital Universitario de Cruces, Barakaldo
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínico de Barcelona, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital San Pedro, Logroño
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta del Hierro, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitari MútuaTerrassa, Terrassa

IPD SHARING:
Plan to Share IPD: Yes
The results will be shared with the investigators involved in the study, and will be shared when the analysis of the results is performed.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months
Access Criteria: Direct collaborators within the study